CLINICAL TRIAL: NCT00379899
Title: A Randomized Study to Evaluate the Effects of Cinacalcet Plus Low Dose Vitamin D on Vascular Calcification in Subjects With Chronic Kidney Disease (CKD) Receiving Hemodialysis
Brief Title: ADVANCE: Study to Evaluate Cinacalcet Plus Low Dose Vitamin D on Vascular Calcification in Subjects With Chronic Kidney Disease Receiving Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060111
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Coronary Artery Calcification; Vascular Calcification; Calcification; Cardiovascular Disease; Chronic Renal Failure; Hyperparathyroidism; Kidney Disease; Nephrology; Secondary Hyperparathyroidism
Keywords: calcification; vascular calcification; coronary vascular calcification; chronic kidney disease; end stage renal disease; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Vascular Calcification; Calcinosis; Cardiovascular Diseases; Hyperparathyroidism; Kidney Diseases; Hyperparathyroidism, Secondary | interventions — Cinacalcet; Vitamin D

ARMS (1):
- Control (Active Comparator): Standard of care, without use of cinacalcet.
  Interventions: Drug: cinacalcet

INTERVENTIONS:
Drug: cinacalcet — Low dose vitamin D with cinacalcet
  Other Names: cinacalcet + low dose vitamin D

SUMMARY:
The purpose of this study is to evaluate whether cinacalcet + low dose vitamin D attenuates the progression of vascular calcification over one year, compared with a treatment regimen that includes flexible vitamin D dosing in the absence of cinacalcet, in subjects with chronic kidney disease receiving hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic kidney disease receiving hemodialysis.
* Lab tests required at screening include Parathyroid Hormone (PTH), calcium, and phosphorus.
* A screening coronary artery calcification score of at least 30.

Exclusion Criteria:

* Subjects on non-calcium or aluminum containing phosphate binders (example: sevelamer HCl, lanthanum) 30 days prior to screening.
* Subjects on cinacalcet 30 days prior to screening.
* Current or previous use of some osteoporosis medications.
* Started or required change in cholesterol lowering medications within 30 days before screening.
* Abnormal rhythm of the heart.
* Parathyroidectomy done within 3 months prior to screening.
* Anticipated parathyroidectomy or kidney transplant.
* Current intolerance to oral medications, or inability to swallow.
* Unstable medical condition.
* Currently enrolled, or fewer than 30 days have passed since subject used another investigational device or drug.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bellasi A, Reiner M, Petavy F, Goodman W, Floege J, Raggi P. Presence of valvular calcification predicts the response to cinacalcet: data from the ADVANCE study. J Heart Valve Dis. 2013 May;22(3):391-9. PMID 24151766
- [Background] Boer R, Lalla AM, Belozeroff V. Cost-effectiveness of cinacalcet in secondary hyperparathyroidism in the United States. J Med Econ. 2012;15(3):509-20. doi: 10.3111/13696998.2012.664799. Epub 2012 Feb 21. PMID 22313328
- [Background] Floege J, Raggi P, Block GA, Torres PU, Csiky B, Naso A, Nossuli K, Moustafa M, Goodman WG, Lopez N, Downey G, Dehmel B, Chertow GM; ADVANCE Study group. Study design and subject baseline characteristics in the ADVANCE Study: effects of cinacalcet on vascular calcification in haemodialysis patients. Nephrol Dial Transplant. 2010 Jun;25(6):1916-23. doi: 10.1093/ndt/gfp762. Epub 2010 Jan 27. PMID 20110249
- [Background] Raggi P, Chertow GM, Torres PU, Csiky B, Naso A, Nossuli K, Moustafa M, Goodman WG, Lopez N, Downey G, Dehmel B, Floege J; ADVANCE Study Group. The ADVANCE study: a randomized study to evaluate the effects of cinacalcet plus low-dose vitamin D on vascular calcification in patients on hemodialysis. Nephrol Dial Transplant. 2011 Apr;26(4):1327-39. doi: 10.1093/ndt/gfq725. Epub 2010 Dec 8. PMID 21148030
- [Background] Urena-Torres PA, Floege J, Hawley CM, Pedagogos E, Goodman WG, Petavy F, Reiner M, Raggi P. Protocol adherence and the progression of cardiovascular calcification in the ADVANCE study. Nephrol Dial Transplant. 2013 Jan;28(1):146-52. doi: 10.1093/ndt/gfs356. Epub 2012 Sep 30. PMID 23028103
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 27 October 2006 through 2 May 2008
Groups:
- Cinacalcet: Cinacalcet plus low dose vitamin D
- Control: Flexible vitamin D dosing
Period: Overall Study
Arm/Group | Cinacalcet | Control
Started | 180 | 180
Completed | 140 | 140
Not Completed | 40 | 40
Not completed — Adverse Event | 7 | 3
Not completed — Death | 10 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 3 | 4
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Ineligibility determined | 0 | 1
Not completed — Noncompliance | 1 | 1
Not completed — Parathyroidectomy | 0 | 2
Not completed — Renal transplantation | 5 | 4
Not completed — Coronary artery bypass graft | 1 | 1
Not completed — Other protocol-specified criteria | 3 | 4
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Control | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (12.6) | 61.8 (12.8) | 61.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 85 | 153
  Male | 112 | 95 | 207
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 6 | 10
  Black or African American | 45 | 40 | 85
  Hispanic or Latino | 11 | 14 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White or Caucasian | 116 | 120 | 236
  Other | 1 | 0 | 1
Coronary Artery Calcification Score Stratification Factor [Number; unit: Participants]
  ≥30 to 399 | 67 | 67 | 134
  ≥400 to 999 | 47 | 47 | 94
  ≥1000 | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in CAC Score
Description: Percent Change from baseline to week 52 in coronary artery calcification (CAC) score. CAC score ranges from 0 to 7500, with 0 representing no calcification.
Time Frame: Baseline and Week 52
Population: Efficacy Evaluable Analysis Set, composed of all randomized participants with a baseline and a week 52 coronary artery calcification score
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Units on a scale | 43.74 (7.40) | 57.39 (7.77)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor (≥ 30 to 399, ≥ 400 to 999, and ≥ 1000)

2. Secondary Outcome: Number of Participants Achieving > 15% Progression of CAC.
Description: Number of participants achieving >15% progression of coronary artery calcification (CAC) at week 52
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Participants | 63 | 77
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.094, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.62, 95% CI [0.36 to 1.08] — Logit estimates (Cinacalcet:Control)

3. Secondary Outcome: Absolute Change in PTH
Description: Absolute change from baseline in intact Parathyroid Hormone (iPTH)
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
pg/mL | -132.86 (29.46) | -71.55 (30.83)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

4. Secondary Outcome: Change From Baseline in AC Score
Description: Change from baseline in aortic calcification (AC) score at week 52. AC score ranges from 0 to >75,000, with 0 representing no calcification.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Units on a scale | 935.92 (233.81) | 1677.28 (385.39)

5. Secondary Outcome: Change From Baseline of the Progression of AVC.
Description: Change from baseline in the aortic valve calcification (AVC) score. AVC score ranges from 0 to >10,000, with 0 representing no calcification.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Units on a scale | 24.29 (24.19) | 55.96 (18.34)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.258, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percent Change in PTH
Description: Percent change from baseline in intact Parathyroid Hormone (iPTH)
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Percentage | -18.18 (5.53) | -3.88 (5.70)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

7. Secondary Outcome: Absolute Change in Calcium
Description: Absolute change from baseline in serum calcium to weeks 44 through 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
mg/dL | -0.51 (0.07) | 0.17 (0.05)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

8. Secondary Outcome: Percent Change in Calcium
Description: Percent change from baseline in corrected serum calcium to weeks 44 through 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Percentage | -5.24 (0.72) | 1.98 (0.59)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

9. Secondary Outcome: Absolute Change in Phosphorus
Description: Absolute change from baseline in serum phosphorus to weeks 44 through 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
mg/dL | -0.92 (0.18) | -0.24 (0.16)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

10. Secondary Outcome: Percent Change in Phosphorus
Description: Percent change from baseline in serum phosphorus to weeks 44 through 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Percentage | -9.63 (2.93) | 5.26 (5.48)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

11. Secondary Outcome: Absolute Change in Ca x P
Description: Absolute change from baseline in corrected serum calcium x phosphorus to week 44 through week 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: (mg/dL)2
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
(mg/dL)2 | -11.22 (1.68) | -1.32 (1.44)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

12. Secondary Outcome: Percent Change in Ca x P
Description: Percent change from baseline in corrected serum calcium x phosphorus (Ca x P) to weeks 44 through 52
Time Frame: Baseline and Weeks 44 through 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Cinacalcet | Control
Number analyzed (Participants) | 115 | 120
Percentage | -14.56 (2.88) | 6.54 (5.15)
Statistical Analysis 1: Comparison: Cinacalcet vs Control; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for screening total coronary artery calcification score stratification factor

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Cinacalcet | Control Group
Serious Adverse Events (participants affected / at risk) | 88/180 | 82/180
Other Adverse Events (participants affected / at risk) | 95/180 | 93/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=180) | Control Group (N=180)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 3
Angina pectoris (Cardiac disorders) | 7 | 4
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 2
Pericardial effusion (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhagic ascites (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 3 | 1
Catheter related complication (General disorders) | 1 | 0
Catheter thrombosis (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Drug intolerance (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 4
Sudden cardiac death (General disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary cyst (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 3 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 3 | 1
Bone abscess (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Catheter related infection (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Central line infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 2 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 2
Localised infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritoneal candidiasis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 7
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 4
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 6 | 3
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 3 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 2 | 3
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 2 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriovenous graft (Surgical and medical procedures) | 1 | 0
Renal transplant (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 2 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 6
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 3 | 3
Labile blood pressure (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 3 | 0
Shock (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=180) | Control Group (N=180)
Anaemia (Blood and lymphatic system disorders) | 6 | 13
Abdominal pain (Gastrointestinal disorders) | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 29 | 22
Nausea (Gastrointestinal disorders) | 29 | 14
Vomiting (Gastrointestinal disorders) | 23 | 22
Chest pain (General disorders) | 5 | 10
Pyrexia (General disorders) | 11 | 13
Nasopharyngitis (Infections and infestations) | 7 | 12
Fall (Injury, poisoning and procedural complications) | 3 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 22
Dizziness (Nervous system disorders) | 10 | 13
Headache (Nervous system disorders) | 13 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Hypertension (Vascular disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.